CLINICAL TRIAL: NCT02295982
Title: Laparoscopic Versus Hand Assisted Laparoscopic Trans-peritoneal Laparoscopic Nephrectomy as One Day Surgery (i.e.: Are There Differences in Postoperative Outcome / Convalescence)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Nessn Azawi, Consultant Urologist, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJ-416
Record Dates: First submitted 2014-11-17; First posted 2014-11-20 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Renal Cancer
Keywords: Laparoscopic nephrectomy; one day surgery
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic nephrectomy (Placebo Comparator): Patient with renal cell carcenoma will undergo laparoscopic nephrectomy within standarized technique
  Interventions: Procedure: Hand assisted laparoscopic nephrectomy
- Hand assisted laparoscopic nephrectomy (Active Comparator): Patient with renal cell carcenoma will undergo hand assisted laparoscopic nephrectomy
  Interventions: Procedure: Hand assisted laparoscopic nephrectomy

INTERVENTIONS:
Procedure: Hand assisted laparoscopic nephrectomy — patients with renal cancer will undergo hans assisted laparoscopic nephrectomy

SUMMARY:
The purpose of this study is to describe the postoperative outcomes after laparoscopic transperitoneal nephrectomy and compare them with hand assisted laparoscopic nephrectomy with a focus on the limiting factors that prevent an ambulatory nephrectomy, and the benefit of our experiences from the previous study to optimize the postoperative outcomes.

ELIGIBILITY:
Inclusion criteria:

1. Patient between 25-80 years old.
2. Diagnosed as Cancer Renis
3. Can read and understand Danish
4. No cardiac disease lead to close cardiologic observations
5. Any T, any N any M stadia.

Exclusion criteria:

1. Mentally sick patient
2. Dement
3. Living alone
4. Cardiac problem
5. Per operative bleeding with the need to blood transfusion
6. Operation time at afternoon

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
postoperative hospital admission | one day

CONTACTS AND LOCATIONS:
Overall Officials: Nessn H Azawi, Principal Investigator — Zealand University Hospital
Locations (1):
- Roskilde Hospital, Roskilde, Denmark